CLINICAL TRIAL: NCT00091910
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of Epoetin Alfa in Critically Ill Subjects
Brief Title: Research Into the Treatment of Anemia for Critically Ill Patients Admitted to Intensive Care Units (ICU)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CR004114
Record Dates: First submitted 2004-09-19; First posted 2004-09-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Anemia
Keywords: Anemia; Epoetin alfa; Erythropoietin; Blood transfusion; Intensive care units
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
Erythropoietin (EPO) is a hormone produced in the kidney. Its function is to stimulate the production of red cells in the bone marrow. The purpose of this research study is to demonstrate that the administration EPO to critically ill subjects in the intensive care unit (ICU) reduces the number of patients requiring red blood cell (RBC) transfusion as compared with placebo (a liquid without active medicine).

DETAILED DESCRIPTION:
In this study the amount of drug and frequency of dosing is under investigation. Erythropoietin (EPO) will be given by subcutaneous injection (a small needle prick placed underneath the skin). The maximum number of injections a patient may receive is 3. The total expected length of time of patient participation in the study is about 140 days (about 5months).

This study consists of a screening period, treatment period and post treatment period. The study doctor will determine whether the patient is suitable for the study. Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures.

Eligible patients will be assigned by chance (like flipping a coin) to one of two treatment groups; 40,000 units of EPO or Placebo. Unless the need arises, neither the patient nor the study staff, will know which treatment the patient receives.

The patient will receive an injection of study drug on Study Days 1, 8 and 15 as long as they remain in the same hospital and their hemoglobin (Hb) level is less than 12g/dL. If the patient's hemoglobin level is greater than 12g/dL on any scheduled medication day, study medication will not be given. However the patient will remain in the study and a re-assessment will be done at the next dosing time point. The patient will also receive iron therapy (at least 150 mg) from Study Day 1 (if tolerated) through Study Day 29 or until the patient is discharge from the hospital or withdraws from the study (whichever comes first).

Treatment with study drug will be stopped if the patient become pregnant, or the study doctor feels that it is in the patient's best interest. If treatment is stopped before Study Day 15, the patient will be required to return for scheduled study assessments through Study Day 140.

The purpose of the post-treatment period is to monitor the patient's health status. Whether or not the patient remains hospitalized, the patient will have two more visits to monitor their health (on Study Day 42 and 140). In addition, the study doctor and nurse will contact the patient or their caregiver by phone monthly following the Study Day 29 visit until Study Day 140. Weekly subcutaneous injections (under the skin) of 40,000 units of EPO or placebo on days 1, 8 and 15.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patient admitted to the ICU
* Patient is anemic when entering the study (hemoglobin </= 12.0 g/dL)

Exclusion Criteria:

* Patients with a history of blood clots (deep vein thrombosis)
* Patients with acute ischemic cardiac disease
* Patients receiving hemodialysis or peritoneal dialysis
* Patients admitted to the ICU because of acute GI bleeding
* Patients who are planned to be discharged from the ICU within 48 hours of entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1460 (Actual)
Dates: Start 2003-09; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to demonstrate that the administration of epoetin alfa to critically ill subjects reduces the proportion of subjects requiring red blood cell (RBC) transfusion as compared with placebo at Study Day 29.

SECONDARY OUTCOMES:
Cumulative number of units of red blood cell transfusions received from Study Day 1 through Study Day 42, Change in hemoglobin from Study Day 1 through Study Day 29, Mortality through Study Day 29 and Cumulative mortality through Study Day 140.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Corwin HL, Gettinger A, Fabian TC, May A, Pearl RG, Heard S, An R, Bowers PJ, Burton P, Klausner MA, Corwin MJ; EPO Critical Care Trials Group. Efficacy and safety of epoetin alfa in critically ill patients. N Engl J Med. 2007 Sep 6;357(10):965-76. doi: 10.1056/NEJMoa071533. PMID 17804841
- See also: Research Into the Treatment of Anemia for Critically Ill Patients Admitted to Intensive Care Units (ICU) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=554&filename=CR004114_CSR.pdf